CLINICAL TRIAL: NCT04148586
Title: Randomized Trial Comparing 3 Schedules of Hypofractionated Whole Breast Irradiation in Females With Early Stage Breast Cancer
Brief Title: Trial Comparing 3 Schedules of Hypofractionated Whole Breast Irradiation in Females With Early Stage Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201617090.3
Record Dates: First submitted 2019-02-18; First posted 2019-11-01 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- One week Whole Breast Irradiation (Experimental): WBI: 27 Gy/5 fractions/1 week. 5.4 Gy /fraction ± boost to tumor bed 5.4 Gy/ 1 fraction, 2 days after the end of WBI.
  Interventions: Other: Whole Breast Irradiation
- Once weekly Whole Breast Irradiation (Experimental): WBI: 28.5 Gy/ 5 fractions/ 5 weeks. 5.7 Gy/fraction ± boost to tumor bed 5.7 Gy/ 1 fraction, one week after the end of WBI. WBI is given on the same day each week.
  Interventions: Other: Whole Breast Irradiation
- 3 weeks Whole Breast Irradiation (Active Comparator): WBI: 40.05 Gy/ 15 fractions/ 3 weeks. 2.67 Gy/ fraction ± boost to tumor bed 10 Gy/ 4 fraction / 4 days after the end of WBI
  Interventions: Other: Whole Breast Irradiation

INTERVENTIONS:
Other: Whole Breast Irradiation — Whole Breast Irradiation after CBS in females with DCIS and early stage breast cancer

SUMMARY:
The establishment of conservative breast surgery (CBS) and whole breast irradiation (WBI) as an alternative to mastectomy was a process that occurred over two to three decades. Based on the available evidence, hypofractionated WBI may be safely offered to most women with ductal carcinoma insitu (DCIS) or early-stage invasive breast cancer after CBS. This prospective randomized clinical trial aims to evaluate the outcomes of one-week and once weekly schedules of WBI against the investigator's standard hypofractionated WBI ( 40 Gy /15 fraction /3 weeks) in females with early stage breast cancer after CBS.

DETAILED DESCRIPTION:
1. Radiotherapy Timing If the patient is not receiving chemotherapy, WBI is to be initiated within 9 weeks following lumpectomy or re-excision of margins. For patients receiving chemotherapy, WBI is to begin no fewer than 2 weeks and no more than 8 weeks after the last cycle of chemotherapy.
2. Randomization:

138 patients will be randomized using permuted blocks randomization to 3 equal comparable arms.

- Dose Prescriptions

Arm 1:

One week WBI: 27Gy/5 fractions /1 week. 5.4 Gy/fraction ± boost to tumor bed 5.4 Gy/ 1 fraction, 2 days after the end of WBI.

Arm 2:

Once weekly WBI: 28.5 Gy/ 5 fractions/ 5 weeks. 5.7 Gy/fraction ± boost to tumor bed 5.7 Gy/ 1 fraction, one week after the end of WBI. WBI is given on the same day each week.

Arm 3:

Hypofractionated WBI 40 Gy/ 15 fractions/ 3 weeks. 2.67 Gy/ fraction ± boost to tumor bed 10 Gy/ 4 fraction / 4 days after the end of WBI.

3-Tumor bed boost A tumor bed boost is recommended to high-risk patients [Age < 50 years, high grade] according to the National Comprehensive Cancer Network (NCCN) guidelines.

4-Radiotherapy simulation, Localization and Outlining:

* The guidelines for contouring will conform to the policies set by the Radiation Therapy Oncology Group (RTOG) Breast cancer Atlas. www.rtog.org/CoreLab/ContouringAtlases/BreastCancerAtlas.aspx
* Megavoltage ( MV) photon beams with energies ≥ 6 MV are required.
* Radiotherapy Planning:

Computed tomography based conformal radiotherapy (CT-based 3D-CRT) planning with tissue inhomogeneity correction is required .

5- Systemic Therapy

* Chemotherapy Adjuvant chemotherapy may be given at the discretion of the patient's medical oncologist. The use of chemotherapeutic agents during radiation therapy is not allowed. The use of neoadjuvant chemotherapy is not allowed.
* Hormonal therapy Patients with ER-positive and/or PR-positive tumors should be treated with hormonal therapy for a minimum of 5 years. The use of hormonal therapy during radiation therapy is allowed.
* Trastuzumab Trastuzumab is given to HER2 positive patients. The use of Trastuzumab during radiation therapy is allowed.

  6-Surgical Treatment:
* All patients will undergo CBS, axillary staging and/or dissection with negative surgical margins (sm).
* Negative surgical margin (Curigliano, 2017)

  * Invasive breast cancer: no ink on tumor
  * DCIS: 2mm
* Surgical clips will be used to define the tumor bed borders
* Breast reconstruction and cosmetic breast implants are not allowed 7-Follow-up.

Schedule of Follow up:

* History and physical exam for all randomized patients will occur every 3 months in the first 2 years after the date of end of radiotherapy treatment
* Monitor and refer for lymphedema management.
* Mammography will be requested annually

ELIGIBILITY:
Inclusion Criteria:

* Tis, pT1-2, pN0-1, M0 disease
* Invasive carcinoma of the breast or ductal carcinoma insitu [DCIS]
* CBS (reconstruction is not allowed)
* Negative surgical margin
* Axillary staging &/or dissection

Exclusion Criteria:

* pT3-4, pN2-3 breast cancer
* Inadequate axillary lymph node dissection
* Neoadjuvant chemotherapy
* Non-epithelial breast malignancies such as sarcoma or lymphoma
* Synchronous bilateral invasive or non-invasive breast cancer
* History of invasive breast cancer or DCIS (Patients with a history of lobular carcinoma in situ (LCIS) treated by surgery alone are eligible.)
* Past history of malignancy except
* Basal cell skin cancer
* CIN cervix uteri
* Cosmetic breast implants (Patients who have had implants removed are eligible.)
* Prior breast or thoracic RT for any condition
* Collagen vascular disease, specifically systemic lupus, or scleroderma
* Pregnancy or lactation at the time of radiotherapy. Women of reproductive potential must agree to use an effective non-hormonal method of contraception during therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Acute toxicity | 3 months from the start of whole breast irradiation
  The proportion of patients with grade ≥3 toxicity according to The Radiation Therapy Oncology Group (RTOG) morbidity scoring criteria.
Cosmetic outcome | Annually after the end of whole breast irradiation for 5 years
  measured by The European Organisation for Research and Treatment of Cancer (EORTC) breast cosmetic rating system (observer rating)
Ibsilateral locoregional tumor control | Annually after the end of whole breast irradiation for 5 years.
  must be confirmed by cytological/ histological assessment
patient-reported outcome measures (PROMs) | Annually after the end of whole breast irradiation for 5 years.
  measured by The European Organisation for Research and Treatment of Cancer, EORTC Quality of Life questionnaire for breast cancer patients ( EORTC QLQ-BR 23).

SECONDARY OUTCOMES:
late toxicity | Annually after the end of whole breast irradiation for 5 years.
  Late toxicity according to The Radiation Therapy Oncology Group/ The European Organisation for Research and Treatment of Cancer (RTOG/EORTC) late radiation morbidity scoring schema
Distant disease-free survival | 5 years from the initial diagnosis of breast cancer
  Defined as the time from initial diagnosis of breast cancer to first diagnosis of distant disease, regardless of the occurrence of any intervening local or regional failure, contralateral breast cancer, or non-breast second primary cancer.
Overall survival | 5 years from the initial diagnosis of breast cancer
  Defined as the time from initial diagnosis of breast cancer to date of death or last follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Marwa M El Awadly, Principal Investigator — National Cancer Institute, Cairo University, Egypt
Locations (1):
- NCI. Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Sharing plan includes study protocol, statistical analysis plan, informed consent form and clinical study report.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: January 2021
Access Criteria: marwa.awadly@nci.cu.edu.eg

REFERENCES:
- [Result] Brunt AM, Wheatley D, Yarnold J, Somaiah N, Kelly S, Harnett A, Coles C, Goodman A, Bahl A, Churn M, Zotova R, Sydenham M, Griffin CL, Morden JP, Bliss JM; FAST-Forward Trial Management Group. Acute skin toxicity associated with a 1-week schedule of whole breast radiotherapy compared with a standard 3-week regimen delivered in the UK FAST-Forward Trial. Radiother Oncol. 2016 Jul;120(1):114-8. doi: 10.1016/j.radonc.2016.02.027. Epub 2016 Apr 1. PMID 27046390
- [Result] • Fast forward protocol, Version 3.0: 08/07/2015: https://njl-admin.nihr.ac.uk/document/download/2006786.
- [Result] FAST Trialists group; Agrawal RK, Alhasso A, Barrett-Lee PJ, Bliss JM, Bliss P, Bloomfield D, Bowen J, Brunt AM, Donovan E, Emson M, Goodman A, Harnett A, Haviland JS, Kaggwa R, Morden JP, Robinson A, Simmons S, Stewart A, Sydenham MA, Syndikus I, Tremlett J, Tsang Y, Wheatley D, Venables K, Yarnold JR. First results of the randomised UK FAST Trial of radiotherapy hypofractionation for treatment of early breast cancer (CRUKE/04/015). Radiother Oncol. 2011 Jul;100(1):93-100. doi: 10.1016/j.radonc.2011.06.026. PMID 21752481
- [Result] Haviland JS, Owen JR, Dewar JA, Agrawal RK, Barrett J, Barrett-Lee PJ, Dobbs HJ, Hopwood P, Lawton PA, Magee BJ, Mills J, Simmons S, Sydenham MA, Venables K, Bliss JM, Yarnold JR; START Trialists' Group. The UK Standardisation of Breast Radiotherapy (START) trials of radiotherapy hypofractionation for treatment of early breast cancer: 10-year follow-up results of two randomised controlled trials. Lancet Oncol. 2013 Oct;14(11):1086-1094. doi: 10.1016/S1470-2045(13)70386-3. Epub 2013 Sep 19. PMID 24055415
- [Result] Dragun AE, Ajkay NJ, Riley EC, Roberts TL, Pan J, Rai SN, Jain D, Quillo AR, Scoggins CR, McMasters KM, Woo SY. First Results of a Phase 2 Trial of Once-Weekly Hypofractionated Breast Irradiation (WHBI) for Early-Stage Breast Cancer. Int J Radiat Oncol Biol Phys. 2017 Jul 1;98(3):595-602. doi: 10.1016/j.ijrobp.2017.01.212. PMID 28581400